CLINICAL TRIAL: NCT00445432
Title: A Multi-Center, Randomized, Double-blind, Placebo-controlled Study of Adalimumab for the Maintenance of Clinical Remission in Japanese Subjects With Crohn's Disease
Brief Title: A Study of Adalimumab for the Maintenance of Clinical Remission in Japanese Subjects With Crohn's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-837
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- DB Adalimumab 40 mg eow (Experimental): Subjects received double-blind (DB) 40 mg adalimumab subcutaneously (SC) every other week (eow) during the DB treatment period lasting 52 weeks.
  Interventions: Biological: adalimumab
- Placebo eow (Placebo Comparator): Subjects received placebo subcutaneously (SC) every other week (eow) during the double-blind treatment period lasting 52 weeks.
  Interventions: Other: Placebo
- OL Adalimumab 40 mg eow (Experimental): Subjects received open-label (OL) 40 mg adalimumab subcutaneously (SC) every other week (eow) during the double-blind treatment period lasting 52 weeks.
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — Subcutaneous injection of 40 mg adalimumab (0.8 mL/injection) every other week (eow)
  Other Names: Humira; D2E7
  Arms: DB Adalimumab 40 mg eow; OL Adalimumab 40 mg eow
Other: Placebo — Subcutaneous injection of placebo (0.8 mL/injection) every other week (eow)
  Arms: Placebo eow

SUMMARY:
To demonstrate the efficacy and safety of adalimumab for the maintenance of clinical remission in Japanese subjects with Crohn's disease.

DETAILED DESCRIPTION:
This was a Phase 2/3, multicenter, randomized, double-blind (DB), placebo-controlled, two-arm, efficacy, safety, and pharmacokinetic study designed to demonstrate the effectiveness of adalimumab in Japanese patients with moderate to severe Crohn's Disease (CD).

All participants who had completed Study M04-729 (NCT00445939), the lead-in adalimumab induction therapy study, were eligible for this study. Participants who rolled over into this study received either DB treatment (adalimumab or placebo) or open-label (OL) treatment with adalimumab.

Crohn's Disease Activity Index (CDAI) was used to determine participants who were responders and participants who were in clinical remission. CDAI documents number of soft stools, abdominal pain, general well-being, presence of 6 signs (arthritis/arthralgia; iritis/uveitis; erythema nodosum/pyoderma gangrenosum/aphthous stomatitis; fissure, abscess, anal fistula; other cutaneous fistula; fever over 100 degrees), taking medication for diarrhea, abdominal mass, hematocrit, and weight loss during a 1-week assessment period. It yields a total score >= 0 and without upper limit. Baseline scores in the study ranged from 221 to 448. Low score=less severe CD activity. Decrease in score indicates improvement.

Clinical remission is a CDAI score < 150.

Clinical response-70 (CR-70) = decrease in CDAI ≥ 70 points from lead-in study Baseline score.

Clinical response-100 (CR-100) = decrease in CDAI ≥ 100 points from lead-in study Baseline score.

Participants who had CR-70 response at Week 4 of the induction study were randomized into 1 of 2 treatment groups (double-blind adalimumab 40 mg every other week or adalimumab placebo every other week) using 2 stratification factors - CDAI category (CDAI less than 150 and CDAI 150 or higher) and presence/absence of fistula at Week 0 of this study. The double-blind treatment was to last from Week 0 to Week 52. Any time at or after Week 4 of this study, if a participant's disease flared (defined as a recurrence of very active disease, specifically an increase in CDAI when compared to Week 0 in this study of ≥ 70 points and a CDAI above 220) during the double-blind treatment period, the participant was allowed to move to OL treatment. At Week 52, all participants still receiving DB treatment were to be moved to open-label treatment and could continue in the study until adalimumab is approved for commercial use in Japan.

Participants who did not respond by Week 4 in the induction study and participants who had disease flare during DB treatment of this study entered OL treatment and received adalimumab 40 mg every other week. At or after Week 4 of this study, if a participant in the open-label treatment group had a disease flare or if the participant was still not responding to treatment, the participant was allowed to dose escalate to adalimumab 80 mg every other week. Participants who entered open-label treatment were to be allowed to continue on open-label adalimumab until adalimumab is approved for commercial use in Japan.

The study is complete. Results of this study are reported for endpoints at Week 52 (end of the DB treatment period) for subjects who received DB treatment (adalimumab or placebo) or OL adalimumab treatment and for endpoints at Week 148 for all subjects who received at least one dose of adalimumab in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who successfully enrolled in and completed the M04-729, (NCT00445939) study

Exclusion Criteria:

* Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Kobayashi, Study Director — Abbott
Locations (29):
- Japan (29):
  - Site Ref # / Investigator 46965, Aichi
  - Site Ref # / Investigator 46977, Aichi
  - Site Ref # / Investigator 46978, Aichi
  - Site Ref # / Investigator 46979, Aichi
  - Site Ref # / Investigator 46922, Chiba
  - Site Ref # / Investigator 46974, Chiba
  - Site Ref # / Investigator 46970, Ehime
  - Site Ref # / Investigator 46971, Fukuoka
  - Site Ref # / Investigator 46985, Fukuoka
  - Site Ref # / Investigator 46986, Fukuoka
  - Site Ref # / Investigator 46987, Fukuoka
  - Site Ref # / Investigator 46968, Hiroshima
  - Site Ref # / Investigator 46973, Hokkaido
  - Site Ref # / Investigator 6881, Hokkaido
  - Site Ref # / Investigator 46982, Hyōgo
  - Site Ref # / Investigator 46969, Kagawa
  - Site Ref # / Investigator 46927, Kanagawa
  - Site Ref # / Investigator 46984, Kochi
  - Site Ref # / Investigator 46981, Kyoto
  - Site Ref # / Investigator 46921, Miyagi
  - Site Ref # / Investigator 46983, Okayama
  - Site Ref # / Investigator 46966, Osaka
  - Site Ref # / Investigator 46967, Osaka
  - Site Ref # / Investigator 46980, Shiga
  - Site Ref # / Investigator 46964, Shizuoka
  - Site Ref # / Investigator 46923, Tokyo
  - Site Ref # / Investigator 46924, Tokyo
  - Site Ref # / Investigator 46975, Tokyo
  - Site Ref # / Investigator 46976, Tokyo

REFERENCES:
- [Derived] Watanabe M, Hibi T, Mostafa NM, Chao J, Arora V, Camez A, Petersson J, Thakkar R. Long-term safety and efficacy of adalimumab in Japanese patients with moderate to severe Crohn's disease. J Crohns Colitis. 2014 Nov;8(11):1407-16. doi: 10.1016/j.crohns.2014.04.012. Epub 2014 May 27. PMID 24874893
- [Derived] Watanabe M, Hibi T, Lomax KG, Paulson SK, Chao J, Alam MS, Camez A; Study Investigators. Adalimumab for the induction and maintenance of clinical remission in Japanese patients with Crohn's disease. J Crohns Colitis. 2012 Mar;6(2):160-73. doi: 10.1016/j.crohns.2011.07.013. Epub 2011 Aug 26. PMID 22325170

RESULTS

PARTICIPANT FLOW:
Groups:
- DB Adalimumab 40 mg Eow: Double-blind adalimumab 40 mg every other week
- Placebo Eow: Double-blind adalimumab placebo every other week
- OL Adalimumab 40 mg Eow: Open-label adalimumab 40 mg every other week
- Any Adalimumab: All participants in NCT00445432 (Study M06-837) who received at least 1 dose of adalimumab 40 mg every other week (double-blind or open-label).
Period: Through Week 52 of NCT00445432 (M06-837)
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow | OL Adalimumab 40 mg Eow | Any Adalimumab
Started | 25 | 25 | 32 | 0 (This treatment group is not applicable for this period.)
Completed | 10 | 2 | 21 | 0
Not Completed | 15 | 23 | 11 | 0
Not completed — Adverse Event | 1 | 2 | 7 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Moved to open-label | 14 | 20 | 0 | 0
Not completed — Other | 0 | 1 | 2 | 0
Period: 148 Weeks of Adalimumab Treatment
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow | OL Adalimumab 40 mg Eow | Any Adalimumab
Started | 0 (This group is not applicable for this period.) | 0 (This group is not applicable for this period.) | 0 (This group is not applicable for this period.) | 79 (3 participants discontinued while receiving double-blind placebo and never received any adalimumab)
Completed | 0 | 0 | 0 | 35
Not Completed | 0 | 0 | 0 | 44
Not completed — Adverse Event | 0 | 0 | 0 | 32
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow | OL Adalimumab 40 mg Eow | Total
Number analyzed (Participants) | 25 | 25 | 32 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 3 | 5
  Between 18 and 65 years | 25 | 23 | 29 | 77
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.60 (7.171) | 30.80 (10.939) | 30.75 (8.359) | 31.02 (8.808)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 14 | 33
  Male | 16 | 15 | 18 | 49
Region of Enrollment [Number; unit: participants]
  Japan | 25 | 25 | 32 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Clinical Remission at Week 52 of Double-blind Treatment
Description: Clinical remission=Crohn's Disease (CD) Activity Index (CDAI) <150; number of soft stools, abdominal pain, general well-being, presence of 6 signs (arthritis/arthralgia; iritis/uveitis; erythema nodosum/pyoderma gangrenosum/aphthous stomatitis; fissure, abscess, anal fistula; other cutaneous fistula; fever over 100 degrees), taking medication for diarrhea, abdominal mass, hematocrit, and weight loss are documented during 1-week assessment period. CDAI total score is >= 0 and without upper limit. Low score=less severe CD activity. Decrease indicates improvement.
Time Frame: Week 52 of double-blind treatment
Population: Modified Full Analysis Set (mFAS), defined as participants who had received adalimumab (not placebo) during the adalimumab induction study and who received at least 1 dose of DB study drug during this study. Nonresponder imputation (NRI) (clinical remission not achieved) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow
Number analyzed (Participants) | 21 | 22
Participants | 8 | 2

2. Secondary Outcome: Number of Participants Who Had Clinical Response-70 (CR-70; a Decrease in Crohn's Disease Activity Index of at Least 70 Points From Lead-in Study [NCT00445939] Baseline Score) at Week 52 of Double-blind Treatment
Description: Crohn's Disease Activity Index (CDAI) documents number of soft stools, abdominal pain, general well-being, presence of 6 signs (arthritis/arthralgia; iritis/uveitis; erythema nodosum/pyoderma gangrenosum/aphthous stomatitis; fissure, abscess, anal fistula; other cutaneous fistula; fever over 100 degrees), taking medication for diarrhea, abdominal mass, hematocrit, and weight loss during a 1-week assessment period. CDAI has a total score >= 0 and without upper limit. Low score=less severe CD activity. Decrease in score indicates improvement.
Time Frame: Week 52 of double-blind treatment
Population: OL efficacy set (assigned to OL treatment at Week 0, received >= 1 dose of OL study drug) and mFAS (participants who had received adalimumab [not placebo] during adalimumab induction study and who received >= 1 dose of DB study drug during this study). Nonresponder imputation (NRI) (CR-70 not achieved) used for DB treatments; LOCF for OL treatment.
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 21 | 22 | 32
Participants | 9 | 2 | 10

3. Secondary Outcome: Number of Participants Who Had Clinical Response-100 (CR-100; a Decrease in Crohn's Disease Activity Index of at Least 100 Points From Lead-in Study [NCT00445939] Baseline Score) at Week 52 of Double-blind Treatment
Description: as for outcome 2
Time Frame: Week 52 of double-blind treatment
Population: OL efficacy set (assigned to OL treatment at Week 0, received >= 1 dose of OL study drug) and mFAS (participants who had received adalimumab (not placebo) during adalimumab induction study and who received >= 1 dose of DB study drug during this study). NRI (CR-100 not achieved) used for missing data for DB treatments; LOCF for OL treatment.
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 21 | 22 | 32
Participants | 8 | 2 | 8

4. Secondary Outcome: Change in Crohn's Disease Activity Index From Baseline of Lead-in Study (NCT00445939) to Week 52 of Double-blind Treatment
Description: Crohn's Disease Activity Index (CDAI) is a measure of disease severity. Number of soft stools, abdominal pain, general well-being, presence of 6 signs (arthritis/arthralgia; iritis/uveitis; erythema nodosum/pyoderma gangrenosum/aphthous stomatitis; fissure, abscess, anal fistula; other cutaneous fistula; fever over 100 degrees), taking medication for diarrhea, abdominal mass, hematocrit, and weight loss are documented during 1-week assessment period. CDAI has a total score >= 0 and without upper limit. Low score=less severe CD activity. Decrease in score indicates improvement.
Time Frame: Baseline of lead-in study (NCT00445939) to Week 52 of double-blind treatment
Population: modified Full Analysis Set (mFAS), defined as participants who had received adalimumab (not placebo) during the adalimumab induction study and who received at least 1 dose of DB study drug during this study. Last observation carried forward (LOCF) used for missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow
Number analyzed (Participants) | 21 | 22
units on a scale | -83.7 (110.26) | -9.1 (110.41)

5. Secondary Outcome: Number of Participants Who Had Clinical Remission at Week 52 of Open-label Treatment
Description: Clinical remission=Crohn's Disease (CD) Activity Index (CDAI) <150; number of soft stools, abdominal pain, general well-being, presence of 6 signs (arthritis/arthralgia; iritis/uveitis; erythema nodosum/pyoderma gangrenosum/aphthous stomatitis; fissure, abscess, anal fistula; other cutaneous fistula; fever over 100 degrees), taking medication for diarrhea, abdominal mass, hematocrit, and weight loss are documented during 1-week assessment period. CDAI total score is >= 0 and without upper limit. Low score=less severe CD activity. Decrease in score indicates improvement.
Time Frame: Week 52 of open-label treatment
Population: OL efficacy set (assigned to OL treatment at Week 0, received >= 1 dose of OL study drug). Last observation carried forward (LOCF) used for missing data.
Measure: Number; unit: Participants
Arm/Group | OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 32
Participants | 5

6. Secondary Outcome: Change in International Organization for the Study of Inflammatory Bowel Disease (IOIBD) Score From Baseline of Lead-in Study (NCT00445939) to Week 52 of Double-blind Treatment
Description: The International Organization for the Study of Inflammatory Bowel Disease (IOIBD) score is an indicator of the activity of Crohn's disease. It measures absence (score of 0) or presence (score of 1) of abdominal pain, diarrhea or bloody stools more than 6 times per day, anal lesion, anal fistula, other complication, abdominal mass, weight loss, fever above 38 degrees Centigrade, abdominal tenderness, and blood pigment below 10 g/dL. Total possible score=0 to 10; low score=less disease activity. Decrease in score indicates alleviation of the disease; increase indicates aggravation of disease.
Time Frame: Baseline of lead-in study (NCT00445939) to Week 52 of double-blind treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow
Number analyzed (Participants) | 21 | 22
units on a scale | -0.8 (1.89) | -0.2 (1.34)

7. Secondary Outcome: Change in Inflammatory Bowel Disease Questionnaire (IBDQ) From Baseline of Lead-in Study (NCT00445939) to Week 52 of Double-blind Treatment
Description: IBDQ is a validated disease-specific instrument that assesses the impact of IBD on patient quality of life during a 2-week recall period. It has 32 questions about bowel function and related symptoms, and their social and emotional impact. For each item, participants select 1 of 7 responses. 1=poor quality of life (e.g., feeling of fatigue "all of the time") and 7=good quality (e.g., feeling of fatigue "none of the time"). Scoring range = 32 to 224. Higher scores indicate better quality of life; increases in IBDQ = improved overall quality of life.
Time Frame: Baseline of lead-in study (NCT00445939) to Week 52 of double-blind treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow
Number analyzed (Participants) | 16 | 14
units on a scale | 27.8 (32.44) | 1.8 (35.42)

8. Secondary Outcome: Change in Physical Component of the Short Form-36 Health Survey From Baseline of the Lead-in Study (NCT00445939) to Week 52 of Double-blind Treatment
Description: The Short-Form-36 (SF-36) Health Survey is a comprehensive quality of life scale. An increase in SF-36 score indicates alleviation of the disease and a decrease in score indicates aggravation of disease. The physical component reflects activity level, activity limitations, pain, and rating of one's health. Score on the physical component ranges from 0 (Poorest Health) to 100 (Best Health).
Time Frame: Baseline of lead-in study (NCT00445939) to Week 52 of double-blind treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow
Number analyzed (Participants) | 16 | 14
units on a scale | 4.4 (9.09) | 0.2 (6.31)

9. Secondary Outcome: Change in Mental Component of the Short Form-36 Health Survey From Baseline of the Lead-in Study (NCT00445939) to Week 52 of Double-blind Treatment
Description: The Short-Form-36 (SF-36) Health Survey is a comprehensive quality of life scale. An increase in SF-36 score indicates alleviation of the disease and a decrease in score indicates aggravation. The mental component reflects energy/vitality, social functioning, limitations, and ratings of one's mental health. Score on mental component ranges from 0 (worst score) to 100 (best score).
Time Frame: Baseline of lead-in study (NCT00445939) to Week 52 of double-blind treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow
Number analyzed (Participants) | 16 | 14
units on a scale | 9.6 (8.37) | 0.3 (14.15)

10. Other Pre Specified Outcome: Number of Participants Who Had Clinical Remission at Week 148
Description: Clinical remission = Crohn's Disease (CD) Activity Index (CDAI) <150; number of soft stools, abdominal pain, general well-being, presence of 6 signs (arthritis/arthralgia; iritis/uveitis; erythema nodosum/pyoderma gangrenosum/aphthous stomatitis; fissure, abscess, anal fistula; other cutaneous fistula; fever over 100 degrees), taking medication for diarrhea, abdominal mass, hematocrit, and weight loss are documented during 1-week assessment period. CDAI total score is >= 0 and without upper limit. Low score=less severe CD activity. Decrease indicates improvement.
Time Frame: Week 148 relative to the first dose of adalimumab in NCT00445432 (Study M06-837)
Population: Data is reported as observed cases. No imputation technique was used.
Measure: Number; unit: participants
Groups:
- Any Adalimumab: All participants in this study who received at least 1 dose of adalimumab 40 mg every other week (double-blind or open-label).
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 36
participants | 21

11. Other Pre Specified Outcome: Number of Participants Who Had Clinical Response-70 (CR-70; a Decrease in Crohn's Disease Activity Index of at Least 70 Points From Lead-in Study [NCT00445939] Baseline Score) at Week 148
Description: as for outcome 2
Time Frame: Week 148 relative to the first dose of adalimumab in NCT00445432 (Study M06-837)
Population: Data is reported as observed cases. No imputation technique was used.
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 36
participants | 28

12. Other Pre Specified Outcome: Number of Participants Who Had Clinical Response-100 (CR-100; a Decrease in Crohn's Disease Activity Index of at Least 100 Points From Lead-in Study [NCT00445939] Baseline Score) at Week 148
Description: as for outcome 2
Time Frame: Week 148 relative to the first dose of adalimumab in NCT00445432 (Study M06-837)
Population: Data is reported as observed cases. No imputation technique was used.
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 36
participants | 26

13. Other Pre Specified Outcome: Change in Crohn's Disease Activity Index From Baseline of Lead-in Study (NCT00445939) to Week 148
Description: Crohn's Disease Activity Index (CDAI) is a measure of disease severity. Number of soft stools, abdominal pain, general well-being, presence of 6 signs (arthritis/arthralgia; iritis/uveitis; erythema nodosum/pyoderma gangrenosum/apthous stomatitis; fissure, abscess, anal fistula; other cutaneous fistula; fever over 100 degrees), taking medication for diarrhea, abdominal mass, hematocrit, and weight loss are documented during 1-week assessment period. CDAI has a total score >=0 and without upper limit. Low score=less severe CD activity. Decrease in score indicates improvement.
Time Frame: Baseline of lead-in study (NCT00445939) to Week 148 relative to the first dose of adalimumab in NCT00445432 (Study M06-837)
Population: Data is reported as observed cases. No imputation technique was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 36
units on a scale | -143.0 (102.49)

14. Other Pre Specified Outcome: Change in International Organization for the Study of Inflammatory Bowel Disease (IOIBD) Score From Baseline of Lead-in Study (NCT00445939) to Week 148
Description: as for outcome 6
Time Frame: as for outcome 13
Population: Data is reported as observed cases. No imputation technique was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 35
units on a scale | -1.7 (1.41)

15. Other Pre Specified Outcome: Change in Inflammatory Bowel Disease Questionnaire (IBDQ) From Baseline of Lead-in Study (NCT00445939) to Week 148
Description: IBDQ is a validated disease-specific instrument that assesses the impact of IBD on patient quality of life during a 2-week recall period with 32 questions about bowel function and related symptoms & their social/emotional impact. Per item, participants select 1 of 7 responses (1=poor quality of life [e.g., feeling of fatigue "all of the time"]; 7=good quality [e.g., feeling of fatigue "none of the time"]). Scoring range=32 to 224. Higher scores indicate better quality of life; increases in IBDQ=improved overall quality of life.
Time Frame: as for outcome 13
Population: Data is reported as observed cases. No imputation technique was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 37
units on a scale | 27.2 (31.22)

16. Other Pre Specified Outcome: Change in Physical Component of the Short Form-36 Health Survey From Baseline of the Lead-in Study (NCT00445939) to Week 148
Description: The Short Form-36 (SF-36) Health Survey is a comprehensive quality of life scale. An increase in SF-36 score indicates alleviation of the disease and a decrease in score indicates aggravation of disease. The physical component reflects activity level, activity limitations, pain, and rating of one's health. Score on the physical component ranges from 0 to 100, with 0=Poorest Health and 100=Best Health.
Time Frame: as for outcome 13
Population: Data is reported as observed cases. No imputation technique was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 37
units on a scale | 5.44 (7.245)

17. Other Pre Specified Outcome: Change in Mental Component of the Short Form-36 Health Survey From Baseline of the Lead-in Study (NCT00445939) to Week 148
Description: The Short Form-36 (SF-36) Health Survey is a comprehensive quality of life scale. An increase in SF-36 indicates alleviation of the disease and a decrease in score indicates aggravation. The mental component reflects energy/vitality, social functioning, limitations, and ratings of one's mental health. Score on mental component ranges from 0 (worst score) to 100 (best score).
Time Frame: as for outcome 13
Population: Data is reported as observed cases. No imputation technique was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 37
units on a scale | 6.44 (11.173)

ADVERSE EVENTS:
Time Frame: 52 weeks for the double-blind (DB) treatments (adalimumab and placebo) and for the open-label adalimumab treatment. Overall study (maximum adalimumab treatment of 184 weeks plus 70-day follow-up period) for the Any Adalimumab group.
Arm/Group | DB Adalimumab 40 mg Eow | Placebo Eow | OL Adalimumab 40 mg Eow | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 2/25 | 6/25 | 13/32 | 49/79
Other Adverse Events (participants affected / at risk) | 17/25 | 13/25 | 28/32 | 73/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Adalimumab 40 mg Eow (N=25) | Placebo Eow (N=25) | OL Adalimumab 40 mg Eow (N=32) | Any Adalimumab (N=79)
Crohn's disease (Gastrointestinal disorders) | 1 | 3 | 9 | 26
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 4
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0
Perianal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Enterocolitis viral (Infections and infestations) | 0 | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Anal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Large intestinal stricture (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Subdiaphragmatic abscess (Infections and infestations) | 0 | 0 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood phorphorus decreased (Investigations) | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Adalimumab 40 mg Eow (N=25) | Placebo Eow (N=25) | OL Adalimumab 40 mg Eow (N=32) | Any Adalimumab (N=79)
Crohn's disease (Gastrointestinal disorders) | 2 | 4 | 4 | 15
Dental caries (Gastrointestinal disorders) | 3 | 1 | 3 | 16
Adverse drug reaction (General disorders) | 3 | 1 | 6 | 22
Injection site reaction (General disorders) | 2 | 0 | 2 | 6
Pain (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 3 | 17
Nasopharyngitis (Infections and infestations) | 14 | 3 | 23 | 60
Tinea pedis (Infections and infestations) | 2 | 0 | 0 | 0
Antinuclear antibody increased (Investigations) | 2 | 0 | 0 | 7
Blood creatine phosphokinase increased (Investigations) | 1 | 3 | 3 | 6
Headache (Nervous system disorders) | 1 | 2 | 4 | 16
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 6 | 12
Ocular hyperaemia (Eye disorders) | 0 | 0 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Periproctitis (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 2 | 7
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 6
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 11
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 8
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 6
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 9
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 5
Chest pain (General disorders) | 0 | 0 | 0 | 4
Malaise (General disorders) | 0 | 0 | 0 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 4
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 4
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 7
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 4
DNA antibody positive (Investigations) | 0 | 0 | 0 | 5
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 6
Lymphocyte morphology abnormal (Investigations) | 0 | 0 | 0 | 5
Weight decreased (Investigations) | 0 | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 5
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 8
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.